CLINICAL TRIAL: NCT01812005
Title: A Phase II Study of MLN8237 Alone and in Combination With Rituximab in Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphomas
Brief Title: Alisertib With and Without Rituximab in Treating Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow patient enrollment and study discontinued after 14 patients enrolled
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-12106; NCI-2012-02794 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Splenic Marginal Zone Lymphoma; Waldenström Macroglobulinemia
Keywords: MLN8237; B-cell Non Hodgkin Lymphoma; Rituximab
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell | interventions — MLN 8237; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A (alisertib, rituximab) (Experimental): Patients receive alisertib PO BID on days 1-7. Patients unable to achieve CR after course 4 also receive rituximab IV on day 1 of courses 5-12. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: alisertib; Biological: rituximab; Other: laboratory biomarker analysis
- Cohort B (alisertib, rituximab) (Experimental): Patients receive alisertib as in Cohort A. Patients achieving SD or asymptomatic progressive disease after 2 courses also receive rituximab IV on day 1 of courses 3-10. Patients unable to achieve CR by course 4, receive rituximab as in Cohort A. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: alisertib; Biological: rituximab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: alisertib — Given PO
  Other Names: Aurora A kinase inhibitor MLN8237; MLN8237
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Other: laboratory biomarker analysis — Laboratory correlative studies will be performed

SUMMARY:
This phase II trial studies how well alisertib with and without rituximab works in treating patients with relapsed or refractory B-cell non-Hodgkin lymphoma. Alisertib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving alisertib with and without rituximab may be an effective treatment for B-cell non-Hodgkin lymphoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of MLN8237 (alisertib) alone in patients with relapsed and refractory non-Hodgkin lymphoma (NHL) and transformed NHL.

SECONDARY OBJECTIVES:

I. To determine the efficacy of MLN8237 when combined with rituximab in NHL patients who fail to respond to MLN8237 alone in patients with relapsed and refractory NHL and transformed NHL.

II. To determine specific toxicities associated with MLN8237 alone and when combined with rituximab (in NHL patients) in patients with relapsed and refractory NHL and transformed NHL.

III. To determine pharmacokinetics of MLN8237 alone and in combination with rituximab (for NHL patients) in patients with relapsed and refractory NHL and transformed NHL.

IV. To evaluate specific molecular characteristics of the NHL for patients treated with MLN8237 alone and with rituximab in order to correlate particular molecular markers with response and survival.

V. To evaluate long term survival of patients treated with MLN8237 alone and with rituximab.

OUTLINE: Patients are assigned to 1 of 2 treatment groups.

COHORT A: Patients receive alisertib orally (PO) twice daily (BID) on days 1-7. Patients unable to achieve complete response (CR) after course 4 also receive rituximab intravenously (IV) on day 1 of courses 5-12. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

COHORT B: Patients receive alisertib as in Cohort A. Patients achieving stable disease (SD) or asymptomatic progressive disease after 2 courses also receive rituximab IV on day 1 of courses 3-10. Patients unable to achieve CR by course 4, receive rituximab as in Cohort A. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 2 years and then every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically proven relapsed or refractory B-cell NHL of the following World Health Organization (WHO) classification subtypes: follicular lymphoma (FL), mantle cell lymphoma (MCL), lymphoplasmacytic lymphoma/Waldenström's macroglobulinemia (LPL/WM), marginal zone lymphoma (MZL), diffuse large B-cell lymphoma (DLBCL), Burkitt's lymphoma (BL), and B-cell lymphoma with features unclassifiable between Burkitt's and large cell lymphoma; alternatively, patients with histologically proven, newly diagnosed transformed non-Hodgkin's lymphoma (tNHL) are eligible
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* At least one prior therapy; patients with newly diagnosed tNHL are eligible and do not need to have received prior therapy for the transformed lymphoma or prior indolent NHL; prior autologous stem cell transplant is allowed
* Serum creatinine =< 2.0 mg/dL
* Total bilirubin within normal limits
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 1.5 x upper limit of normal
* Absolute neutrophil count (ANC) >= 1000/μL
* Platelet count >= 75,000/μL
* Recovery to =< grade 1 toxicities associated with prior therapy
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study
* Male subject agrees to use an acceptable method for contraception during the entire study treatment period through 4 months after the last dose of MLN8237
* Must be able to take oral medication and to maintain a fast as required for 2 hours before and 1 hour after MLN8237 administration

Exclusion Criteria:

* Pregnant or breast-feeding women and women of childbearing age who are unwilling to use adequate contraception
* Patients with a history of central nervous system involvement by lymphoma
* Patients with known human immunodeficiency virus (HIV), hepatitis B or hepatitis C (active or carriers) are not eligible; this includes all patients with a positive hepatitis C antibody, hepatitis B surface antigen, or hepatitis B core antibody; previously vaccinated patients with positive hepatitis B surface antibody are eligible
* May not have received prior therapy with an Aurora kinase inhibitor
* Patients eligible for and willing to undergo autologous stem cell transplant with curative intent at the time of enrollment are not eligible; patients refractory to at least 2 prior regimens may enroll and proceed to curative autologous transplant if they respond
* Patients who are on chronic steroids for unrelated conditions (i.e. rheumatologic conditions) are not eligible if their total daily dose of steroids is equivalent to greater than 10 mg prednisone
* Radiation therapy to more than 25% of the bone marrow; whole pelvic radiation is considered to be over 25%
* Prior allogeneic bone marrow or organ transplantation
* If applicable, patient has >= grade 2 peripheral neuropathy within 14 days before enrollment
* Known history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease; requirement for supplemental oxygen
* Patients who are on daily proton pump inhibitor therapy must be able to discontinue use or only require use of antacid or hydrogen (H2) antagonist intermittently; patients who require daily administration of proton pump inhibitor, H2 antagonist, or pancreatic enzymes are not eligible; intermittent uses of antacids or H2 antagonists are allowed
* Systemic infection requiring IV antibiotic therapy within 14 days preceding the first dose of study drug, or other severe infection
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities (except asymptomatic patients with a pacemaker with electrocardiogram (ECG) changes reflecting conduction abnormalities secondary to the pacemaker); prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant
* Female subject is pregnant or breast-feeding; confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Other severe acute or chronic medical or psychiatric condition, including uncontrolled diabetes, malabsorption, resection of the pancreas or upper small bowel, requirement for pancreatic enzymes, any condition that would modify small bowel absorption of oral medications, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Treatment with clinically significant enzyme inducers, such as the enzyme- inducing antiepileptic drugs phenytoin, carbamazepine or phenobarbital, or rifampin, rifabutin, rifapentine or St. John's wort within 14 days prior to the first dose of MLN8237 and during the study
* Patients with a corrected QT interval (QTc) at baseline of > 450 milliseconds or other factors that increase the risk of QT prolongation or arrhythmic events (i.e., heart failure, hypokalemia with potassium < 3.5 despite supplementation, family history of long QT syndrome) should be excluded
* Patients who require use of a concomitant medication that can prolong the QT interval and who are unable to discontinue use of this medication during the study period are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-05-21 (Actual); Primary Completion 2015-10-14 (Actual); Study Completion 2017-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Blum, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A (Alisertib, Rituximab) | Cohort B (Alisertib, Rituximab)
Started | 1 | 13
Completed | 1 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Alisertib, Rituximab) | Cohort B (Alisertib, Rituximab) | Total
Number analyzed (Participants) | 1 | 13 | 14
Age, Continuous [Median (Full Range); unit: years] | 77 [77 to 77] | 58 [35 to 73] | 67.5 [35 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 1 | 10 | 11
Region of Enrollment [Number; unit: patients]
  United States | 1 | 13 | 14

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (ORR) to Alisertib Alone
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 18 weeks (6 courses)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort A (Alisertib, Rituximab) | Cohort B (Alisertib, Rituximab)
Number analyzed (Participants) | 1 | 13
percentage of patients | 0 [NA to NA] — 95% Confidence Interval was incalculable due to an insufficient number of events | 15 [2 to 45]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: as for outcome 1
Time Frame: 6 weeks (2 courses)
Population: 2 course endpoints only apply to Cohort B, since Cohort B only received 2 courses of the interested drug
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort A (Alisertib, Rituximab) | Cohort B (Alisertib, Rituximab)
Number analyzed (Participants) | 0 | 13
percentage of patients |  | 8 [0 to 36]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: 95% binomial confidence intervals calculated.
Time Frame: 12 weeks (4 courses)
Population: Data were not collected from the single participant in the "Cohort A (Alisertib, Rituximab)" Arm/Group therfore the 95% Confidence Interval was incalculable due to an insufficient number of events
Arm/Group | Cohort A (Alisertib, Rituximab) | Cohort B (Alisertib, Rituximab)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Response Rate(ORR)
Description: as for outcome 1
Time Frame: 18 weeks (6 courses)
Measure: Number; unit: percentage of patients
Arm/Group | Cohort A (Alisertib, Rituximab) | Cohort B (Alisertib, Rituximab)
Number analyzed (Participants) | 1 | 13
percentage of patients | 0 | 15

5. Secondary Outcome: Complete Response Rate (CR)
Description: as for outcome 1
Time Frame: 6 weeks (2 courses)
Population: 2 course endpoints only apply to Cohort B, since Cohort B only received 2 courses of the interested drug
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort A (Alisertib, Rituximab) | Cohort B (Alisertib, Rituximab)
Number analyzed (Participants) | 0 | 13
percentage of patients |  | 0 [0 to 0]

6. Secondary Outcome: Complete Response Rate
Description: as for outcome 1
Time Frame: 12 weeks (4 courses)
Population: data was not collected for participants in Cohort B (Alisertib, Rituximab)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort A (Alisertib, Rituximab) | Cohort B (Alisertib, Rituximab)
Number analyzed (Participants) | 1 | 0
percentage of patients | NA [NA to NA] — 95% Confidence Interval was incalculable due to an insufficient number of events |

7. Secondary Outcome: Overall Survival
Description: Graphically summarized using the methods of Kaplan and Meier.
Time Frame: Time from study entry to the time of death due to any cause, assessed up to 1 year
Population: data was not collected for participants in Cohort A
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A (Alisertib, Rituximab) | Cohort B (Alisertib, Rituximab)
Number analyzed (Participants) | 0 | 13
months |  | 3.1 [1.7 to 27.6]

8. Secondary Outcome: Progression-free Survival
Description: Graphically summarized using the methods of Kaplan and Meier.
Time Frame: Time from study entry to the time of progression and/or death, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A (Alisertib, Rituximab) | Cohort B (Alisertib, Rituximab)
Number analyzed (Participants) | 1 | 13
months | 2 [NA to NA] — 95% Confidence Interval was incalculable due to an insufficient number of events | 1.2 [.8 to 2.5]

9. Secondary Outcome: Complete Response Rate
Description: as for outcome 1
Time Frame: 18 weeks (6 courses)
Population: The data was not collected and analyzed for this outcome measure
Arm/Group | Cohort A (Alisertib, Rituximab) | Cohort B (Alisertib, Rituximab)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The National Cancer Institutes Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 was used to grade toxicities for patients
Groups:
- Cohort A: Cohort A: Patients receive alisertib PO BID on days 1-7. Patients unable to achieve CR after course 4 also receive rituximab IV on day 1 of courses 5-12. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Cohort B: Cohort B: Patients receive alisertib as in Cohort A. Patients achieving SD or asymptomatic progressive disease after 2 courses also receive rituximab IV on day 1 of courses 3-10. Patients unable to achieve CR by course 4, receive rituximab as in Cohort A. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 0/1 | 10/13
Serious Adverse Events (participants affected / at risk) | 0/1 | 5/13
Other Adverse Events (participants affected / at risk) | 1/1 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=1) | Cohort B (N=13)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) — noninfective
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=1) | Cohort B (N=13)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study had slow patient enrollment and was discontinued after only 14 patients were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes